CLINICAL TRIAL: NCT01087697
Title: A Phase 1 Open Label Exploratory Study of an Autologous Neo-Urinary Conduit in Subjects Requiring Incontinent Urinary Diversion Following Radical Cystectomy
Brief Title: Incontinent Urinary Diversion Using an Autologous Neo-Urinary Conduit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tengion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TNG-CL009
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; radical cystectomy; incontinent urinary diversion
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Implanted with NUC (Experimental): Patients who have been implanted with the Neo-Urinary Conduit
  Interventions: Device: Neo-Urinary Conduit

INTERVENTIONS:
Device: Neo-Urinary Conduit — Implantation with the autologous Neo-Urinary Conduit
  Other Names: NUC

SUMMARY:
The purpose of this study is to see if the Neo-Urinary Conduit(NUC), which is made in the laboratory from a combination of a patient's own cells and other materials can be used to form a conduit to safety allow urine flow from the kidneys to outside the body after radical cystectomy in patients with bladder cancer.

DETAILED DESCRIPTION:
The NUC under investigation is a regenerative medicine product comprised of the patient's own smooth muscle cells, procured from a fat biopsy. Tengion has developed appropriate culture conditions to reproducibly generate the necessary quantities of SMC in vitro from autologous adipose tissue biopsies. The NUC is produced at Tengion's Good Manufacturing Practices (GMP) qualified clinical production facility. In this process, smooth muscle cells (SMC) obtained from an adipose tissue biopsy are propagated ex-vivo for approximately 3 - 4 weeks. At the end of this process, the SMCs are seeded onto the surface of a biodegradable PGA/PLGA mesh scaffold to form the NUC. The NUC is shipped to the investigative site for surgical implantation. Over time, the NUC should facilitate the regeneration of urinary tract tissue.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 18 - 80 years of age
* Patients undergoing radical cystectomy for treatment of bladder cancer clinically staged as no greater than T2, N0
* Indicated and agreed between physician investigator and patient to have an incontinent conduit as the diversion mechanism of choice post cystectomy

Exclusion Criteria:

* History of other cancer within the past 5 years (except non metastatic prostate or non melanoma skin cancer)
* Evidence of cancer metastasis
* History of any pelvic radiation or non-pelvic radiation within past 5 years
* Debilitating cardiac or pulmonary disease
* Expected need for chemotherapy within 3 months post cystectomy
* Life expectancy less than 2 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Structural integrity and conduit patency | 12 months post implantation
  CT scan will be used to demonstrate that urine is able to flow safety through the NUC

SECONDARY OUTCOMES:
Structural integrity and conduit patency | month 12 through month 60 post implantation
  CT scan and renal ultrasound will be used to demonstrate that urine is able to flow safely through the NUC through 60 months post implantation
Procedure and/or product related AEs | month 12 through month 60 post implant
  procedure and/or product related AEs will be evaluated through month 60 post implantation
Overall safety | from enrollment through month 60 post implant
  overall safety will be assess by evaluation of non-product/procedure related adverse events, vital signs and laboratory parameters
Procedure and/or product related adverse events post implantation | through 12 months post implantation
  Evaluation of procedure and/or product related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Gary Steinberg, MD, Principal Investigator — University of Chicago; Trinity J Bivalacqua, M.D., Ph.D., Principal Investigator — The Johns Hopkins Medical Institute
Locations (6):
- United States (6):
  - The University of Chicago, Chicago, Illinois
  - The Johns Hopkins Medical Institutions, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Baylor College of Medicine, Houston, Texas